CLINICAL TRIAL: NCT00927706
Title: Experimental Control Investigation of the Impact of an Assistive Technology Updating and Tune up Intervention on the User-caregiver Dyad: a Multi-site Trial
Brief Title: Experimental Control Investigation of the Impact of Assistive Technology on the User-caregiver Dyad: a Multi-site Trial
Acronym: ATUTI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Responsible Party: Principal Investigator, Louise Demers, Département de l'ergothérapie, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRIUM-8317; NIDRR: H133A060062
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Mobility Limitations
Keywords: Assistive Technology; Mobility Limitation; Physical Disability; Caregiver; Participation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate intervention (Experimental): Subjects and their caregivers randomized to this arm receive the intervention immediately after baseline data is collected.
  Interventions: Device: Assistive technology updating and tune up intervention
- Delayed Intervention (Experimental): Subjects and their caregivers who are randomized to this group will receive the intervention after baseline measurements are administered twice (6 weeks apart).
  Interventions: Device: Assistive technology updating and tune up intervention

INTERVENTIONS:
Device: Assistive technology updating and tune up intervention — This intervention includes 4 components: 1) an in-residence assessment of the mobility preferences of the older person and his/her caregiver; 2) a detailed review of forms of assistance, technological and human, that are currently being used; 3) recommendations by an occupational therapist for possible changes in the older person's mobility assistive technology or assistance strategy; and 4) therapist negotiation of an mobility assistive technology updating and tune-up intervention plan with the individual and his or her caregiver.

SUMMARY:
The purpose of this study is to determine the effectiveness of an assistive technology updating and tune up intervention on users and their caregivers. This intervention includes 4 components:

* an in-residence assessment of the mobility preferences of the older person and his/her caregiver
* a detailed review of forms of assistance, technological and human, that are currently being used
* recommendations by an occupational therapist for possible changes in the older person's mobility assistive technology or assistance strategy
* therapist negotiation of an mobility assistive technology updating and tune-up intervention plan with the individual and his or her caregiver. The intervention is provided to the immediate treatment following the administration of baseline measures and the delayed intervention group six weeks later, after an additional baseline measurement. The treatment is six weeks long and the follow-up is 26 weeks.

Hypothesis 1: For community-dwelling older people, an intervention that increases the appropriateness of existing or new assistive technology(AT) for mobility or self-care will alter established patterns of human assistance, such that caregiver burden is reduced or eliminated.

Hypothesis 2: At the same time, AT users will report less difficulty in mobility or self-care, as well as enhanced subjective well-being, and satisfaction with their modified personal assistance strategy.

Hypothesis 3: Following the AT intervention, caregivers will report reduced physical and/or psychological demands and increased satisfaction with their caregiving-related activities compared with

* the pre-intervention period
* caregivers in a delayed intervention control group. Hypothesis 4: Decreased physical and/or psychological demands on helpers will be associated with increases in device users' satisfaction with their personal assistance strategies.

ELIGIBILITY:
Inclusion Criteria:

* Users: Aged 65 years and over
* Have moderate to severe disability that limits their ability to move from place to place independently and/or to perform self-care activities.
* Living at home
* Receiving 2 or more hour per week of assistance with mobility and/or self-care activities from a non-professional, caregiver who is also willing to take part in the study.
* Those caregivers will be adults aged 18 years and over.

Exclusion Criteria:

* Assistive technology users will be excluded if they have severe aphasia, are currently on a community occupational therapist caseload, or are unable to communicate in English or French.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Life Habits | baseline (1or 2 times), 6 weeks (immediately after intervention), 16 weeks later
Caregivers: Caregiver Assistive Technology Outcome Measure | base line (1 or 2), 6 weeks (immediately after intervention), 16 weeks later

SECONDARY OUTCOMES:
Individually Prioritized Problem Assessment | Baseline (1 or 2 times), Immediately after intervention, 16 weeks later
Functional Autonomy Measurement System | Baseline (1 or 2 times), Immediately after intervention, 16 weeks later
Psychological Impact of Assistive Devices Scale | Imediately after intervention. 16 weeks later
Satisfaction with Personal Assistance Strategy | Baseline (1 or 2 times), Immediately after intervention, 16 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Louise Demers, PhD, Principal Investigator — Université de Montréal
Locations (4):
- Canada (4):
  - Simon Fraser University, Vancovuer, British Columbia
  - Centre de santé et des services sociaux de Bordeaux-Cartierville--St-Laurent, Montreal, Quebec
  - the Centre de santé et des services sociaux Cavendish, Montreal, Quebec
  - the Centre de santé et des services sociaux de Laval, Montreal, Quebec